CLINICAL TRIAL: NCT00972699
Title: Mentor Mothers: A Sustainable Family Intervention in South African Townships
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Human Sciences Research Council (Other Government)
Responsible Party: Principal Investigator, Mary Jane Rotheram-Borus, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01MH077553 (NIH); R01MH077553 (NIH); DAHBR 9A-ASPA
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome; Tuberculosis
Keywords: Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome; Tuberculosis; Women; Pregnancy; Vertical Transmission of Human Immunodeficiency Virus; South Africa; Low Birth Weight
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentor Mothers Intervention (Experimental): In the intervention arm, participants will receive the Department of Health-delivered Prevention of Mother to Child Transmission (PMTCT) program plus the Project Masihambisane mentor mothers support program. HIV positive mentor mothers, who have been through the PMTCT program, will be recruited and trained to deliver the intervention to pregnant mothers living with HIV.
  Interventions: Behavioral: Peer support and mentoring
- Control (No Intervention): Mothers living with HIV in the standard of care control clinics will receive the Department of Health-delivered PMTCT program.

INTERVENTIONS:
Behavioral: Peer support and mentoring — The intervention will be delivered in 4 non consecutive visits during pregnancy and 4 visits post-partum. The sessions will be delivered to mothers living with HIV on the days of their health care appointments either individually or in groups that can accommodate up to 30 mothers living with HIV. The intervention will focus on enhancing the mother-baby relationship through increasing the health of the mother and baby, maintaining the mother's mental health, and reducing HIV transmission.
  Other Names: Masihambisane
  Arms: Mentor Mothers Intervention

SUMMARY:
The purpose of this study is to test a mother-to-mother intervention during pregnancy and after delivery with Mothers Living with HIV (MLH)in South Africa. We hypothesize that the intervention will enhance the adjustment of the children of MLH by improving the health and mental health of MLH which benefits their children, as well as the MLH.

DETAILED DESCRIPTION:
South Africa's HIV/AIDS epidemic, one of the worst in the world, has shown little evidence of decline and is indicative of the urgent need to focus on both preventative and treatment intervention efforts (UNAIDS, 2006). In South Africa, close to one in three women who attend public antenatal clinics are living with HIV (UNAIDS, 2006). In KwaZulu-Natal (KZN) - one of the worst affected provinces - as many as 40% to 60% of pregnant women attending antenatal services are living with HIV (Rochat et al., 2006; Kharsany et al., 2004).

HIV infection in pregnant women raises a number of issues that are not faced by HIV-infected men or non pregnant women (Ojikutu & Stone, 2005) and has particular implications for the successful prevention of mother-to-child transmission (Raisler & Cohn, 2005). Most women learn their HIV status for the first time during antenatal testing, which can be distressing and may introduce or further compound psychological, social and health risks in the antenatal and post natal period (Firn & Norman, 1995; Patel V, Rahman A, Jacob KS, & Hughes M, 2004; Patel, DeSouza, & Rodrigues, 2003; Rochat et al., 2006; Shisana et al., 2005; Stein et al., 2005). Research on the uptake of treatment for HIV indicates that poor mental health and a lack of social support are associated with lowered uptake of HAART (Cook et al., 2006), lowered adherence to anti-retroviral medication (Ammassari, Trotta, Murri, & et al., 2002; DiMatteo, Lepper, & Croghan, 2000; Ickovics et al., 2001; Starace et al., 2002)and increased disease progression (Ickovics et al., 2001).

Fortunately, HIV testing and access to antiretroviral drugs (ARV) to prevent mother-to-child transmission (PMTCT) from HIV positive pregnant women to their babies are currently being scaled up in South Africa (Civil Society HIV and AIDS Congress, 2005; Department of Health, 2005). While the potential exists to cut transmission to babies from mothers living with HIV(MLH), maternal HIV disease has been demonstrated to have negative consequences on maternal mental health and social support and children's emotional, social and developmental outcomes and adjustment - both as a result of chronic HIV illness and as a result of the psychological and social burden of HIV on care giving (Stein et al., 2005; Krebs, Stein, & Rochat, 2005; Stein et al., 2005; Sherr, 2005; Dunn, 2005; Hough, Brumitt, Templin, Saltz, & Mood, 2003).

While PMTCT programs provide the opportunity for women to prevent transmission through medical and feeding interventions, the needs of mothers living with HIV extend well beyond this. The psychosocial challenges facing mothers living with HIV are substantial and, if children are to have positive outcomes, it is necessary to provide mothers living with HIV with the support, skills and knowledge to protect and promote their own health and well-being, that of their babies, and, hopefully, their partners (Rochat et al., 2006; Stein et al., 2005; 2006).

The goal of this randomized trial then is to test an intervention to improve the health and well-being of HIV positive mothers and their babies during pregnancy and the early postpartum period through the implementation of a clinic-based mentor mothers' peer support program(also referred to as Project Masihambisane) and dissemination of health information.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, pregnant, and HIV+
* Enrolled in the PMTCT program at the study site clinic
* Receiving medical care from study site clinic
* Residing in study area for duration of study
* No psychosis, neurological damage, or IQ less than 70, as judged by an interviewer in consultation with a clinical supervisor
* Ability to give informed consent as judged by an interviewer

Exclusion Criteria:

* Less than 18 years, or not pregnant, or not HIV+
* Not enrolled in the PMTCT program at the study site clinic
* Not receiving medical care from study site clinic
* Not residing in study area for duration of study
* Psychosis, neurological damage, or IQ less than 70, as judged by an interviewer in consultation with a clinical supervisor
* Clinical provider (nurse or physician) believes it is not in the best interest of the MLH
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2008-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Baby's health status | 6 days after birth; 6 months after birth; 12 months after birth

SECONDARY OUTCOMES:
Maternal adherence: baby's and mother's health. | 6 days after birth; 6 months after birth; 12 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Rotheram-Borus, Ph.D., Principal Investigator — UCLA Semel Institute, Center for Community Health
Locations (1):
- HSRC Sweetwaters Site, Pietermaritzburg, KwaZulu-Natal, South Africa

REFERENCES:
- [Derived] Christodoulou J, Rotheram-Borus MJ, Bradley AK, Tomlinson M. Home Visiting and Antenatal Depression Affect the Quality of Mother and Child Interactions in South Africa. J Am Acad Child Adolesc Psychiatry. 2019 Dec;58(12):1165-1174. doi: 10.1016/j.jaac.2019.03.016. Epub 2019 Mar 26. PMID 30926571
- [Derived] Rotheram-Borus MJ, Tomlinson M, Roux IL, Stein JA. Alcohol Use, Partner Violence, and Depression: A Cluster Randomized Controlled Trial Among Urban South African Mothers Over 3 Years. Am J Prev Med. 2015 Nov;49(5):715-725. doi: 10.1016/j.amepre.2015.05.004. Epub 2015 Jul 29. PMID 26231855
- [Derived] Richter L, Rotheram-Borus MJ, Van Heerden A, Stein A, Tomlinson M, Harwood JM, Rochat T, Van Rooyen H, Comulada WS, Tang Z. Pregnant women living with HIV (WLH) supported at clinics by peer WLH: a cluster randomized controlled trial. AIDS Behav. 2014 Apr;18(4):706-15. doi: 10.1007/s10461-014-0694-2. PMID 24469222
- [Derived] Rotheram-Borus MJ, Richter LM, van Heerden A, van Rooyen H, Tomlinson M, Harwood JM, Comulada WS, Stein A. A cluster randomized controlled trial evaluating the efficacy of peer mentors to support South African women living with HIV and their infants. PLoS One. 2014 Jan 22;9(1):e84867. doi: 10.1371/journal.pone.0084867. eCollection 2014. PMID 24465444
- [Derived] van Heerden A, Norris S, Tollman S, Richter L, Rotheram-Borus MJ. Collecting maternal health information from HIV-positive pregnant women using mobile phone-assisted face-to-face interviews in Southern Africa. J Med Internet Res. 2013 Jun 10;15(6):e116. doi: 10.2196/jmir.2207. PMID 23748182
- [Derived] Rotheram-Borus MJ, le Roux IM, Tomlinson M, Mbewu N, Comulada WS, le Roux K, Stewart J, O'Connor MJ, Hartley M, Desmond K, Greco E, Worthman CM, Idemundia F, Swendeman D. Philani Plus (+): a Mentor Mother community health worker home visiting program to improve maternal and infants' outcomes. Prev Sci. 2011 Dec;12(4):372-88. doi: 10.1007/s11121-011-0238-1. PMID 21850488
- [Derived] Hartley M, Tomlinson M, Greco E, Comulada WS, Stewart J, le Roux I, Mbewu N, Rotheram-Borus MJ. Depressed mood in pregnancy: prevalence and correlates in two Cape Town peri-urban settlements. Reprod Health. 2011 May 2;8:9. doi: 10.1186/1742-4755-8-9. PMID 21535876
- [Derived] Rotheram-Borus MJ, Richter L, Van Rooyen H, van Heerden A, Tomlinson M, Stein A, Rochat T, de Kadt J, Mtungwa N, Mkhize L, Ndlovu L, Ntombela L, Comulada WS, Desmond KA, Greco E. Project Masihambisane: a cluster randomised controlled trial with peer mentors to improve outcomes for pregnant mothers living with HIV. Trials. 2011 Jan 4;12:2. doi: 10.1186/1745-6215-12-2. PMID 21205302